CLINICAL TRIAL: NCT06825299
Title: Interprofessional Approach to Ultrasound Diagnosis and Intervention in Critical Care Patients With Pneumothorax and/or Hemothorax (Steering the Eagerness Towards Standardization of the Third Core Competency in ICU)
Brief Title: Interprofessional Approach to Ultrasound Diagnosis and Intervention in Critical Care Patients With Pneumothorax and/or Hemothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nader Salama Gaber, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine,Tanta University, Tanta, Egypt., Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36264MS339/9/23
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Interprofessional Approach; Ultrasound; Intervention; Critical Care; Pneumothorax; Hemothorax
MeSH Terms: conditions — Pneumothorax; Hemothorax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group I (Experimental): The Technique was performed according to combination of the BTS guidelines for chest tube insertion and US-guided technique for chest tube insertion by Dev et al. and Menegozzo et al. and US-guided pigtail insertion by Vetrugno et al
  Interventions: Diagnostic Test: Chest-Tube Insertion

INTERVENTIONS:
Diagnostic Test: Chest-Tube Insertion — The technique was performed according to a combination of the Chest-Tube Insertion (BTS) guidelines for chest tube insertion and ultrasound (US)-guided technique for chest tube insertion and US-guided pigtail insertion.

SUMMARY:
Investigate the efficacy of interprofessional team approach to ultrasound guided diagnosis and intervention (pigtail or chest tube insertion) in critical care patients with Pneumothorax and/or hemothorax.

Evaluate the safety of the procedure {Insertion- related complications. Assess the Duration of chest tube insertion

DETAILED DESCRIPTION:
Pneumothorax is defined as the presence of air in the pleural cavity; it can be secondary to underlying pulmonary pathology or trauma. In trauma, about 40-50% of thoracic injuries develop pneumothorax. Traditionally, following the suggestion of the American College of Chest Physicians and the Advanced Trauma Life Support (ATLS), all traumatic pneumothoraxes must be treated with a pleural drainage that could be chest tube (CT) or pigtail catheter (PC).

Insertion of pleural drains is a common surgical procedure. Percutaneous pleural drainage is the third most performed procedure in the intensive care unit (ICU) after vascular catheterization and tracheal intubation.

Bedside-ultrasound is introducing the advantage of at-time diagnosis and evaluation of different parameters without the need for risky transport of critical patients outside ICU and also guiding safe and successful intervention without complications and good learning.

.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 65 years
* Both sexes.
* Patients with pneumothorax or hemothorax indicated for chest tube or pig tail insertion according to British Thoracic Society (BTS) June 2022 guidelines for pleural procedures.

Exclusion Criteria:

* Absolute contraindication: patients in which the lung is completely adherent to the chest wall throughout the hemithorax.
* Relative contraindications: patients with risk of bleeding in patients:
* Taking anticoagulant medication.
* Patients with abnormal clotting profiles, coagulopathies, and platelet defects.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of ultrasound diagnosis | Diagnosis 24 hours
  Efficacy of ultrasound in intervention by Diagnosis of pneumothorax/hemothorax starting by physical examination followed by bed side ultrasound examination according to the international consensus conference recommendations (international evidence-based recommendations for point-of-care lung ultrasound)

SECONDARY OUTCOMES:
Efficacy of ultrasound in intervention | 10 days after intervention
  Efficacy of ultrasound in intervention used (chest tube /pigtail) was recoeded.
Monitoring team performance | 24 hours after intervention
  Monitoring team performance: team satisfaction was recorded using a 5-point Likert scale team satisfaction (1, very dissatisfied; 2, dissatisfied; 3, Okey; 4, satisfied; 5, very satisfied) in our study as an item related to team performance
Duration of insertion | 30 minutes intervention
  Duration of insertion was recorded
Incidence of complications | 72 hours after intervention
  Incidence of complication were recorded such as infection, bleeding, visceral injury, and visceral injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.